CLINICAL TRIAL: NCT01740258
Title: Phase II Trial of Bevacizumab, Radiation Therapy and Temodar Followed by Bevacizumab and Temodar With Continuation of Bevacizumab Beyond Progression (BBP-Bevacizumab Beyond Progression)
Brief Title: Bevacizumab Beyond Progression (BBP)
Acronym: BBP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00038098
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Malignant Glioma; Grade 4 Malignant Glioma; Glioblastoma; Gliosarcoma
Keywords: malignant glioma; Grade 4 malignant glioma; glioblastoma; gliosarcoma; adult brain tumor
MeSH Terms: conditions — Glioma; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Radiotherapy; Temozolomide; norambreinolide-18,6alpha-olide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevaczimab, Radiation Therapy, Temozolomide (Experimental): In Part A, newly-diagnosed patients with Grade 4 malignant gliomas will receive standard radiation therapy, daily Temodar 75mg/M for 6-8 weeks. Bevacizumab will be given concurrently with radiation therapy and Temodar, 10 mg/kg every two weeks.
  If they are stable at the end of Part A, they will continue to Part B. In Part B patients will receive up to 12 cycles of bevacizumab and Temodar. Bevacizumab will be given on Days 1 and 15 of a 28-day cycle. Temodar will be 200 mg/meter squared daily for 5 days (days 1-5) of each cycle.
  If they have not progressed, patients will start Part C. In Part C, patients will receive bevacizumab 10mg/kg approximately every 2 weeks or 15 mg/kg approximately every 3 weeks.
  If patients progress during Part B or C, they will start Part D. In Part D, patients will receive bevacizumab-based therapy containing bevacizumab in combination with a chemotherapy and/or biologic agent, as determined by the Duke treating physician.
  Interventions: Radiation: Radiation Therapy; Drug: Temozolomide; Drug: Bevacizumab

INTERVENTIONS:
Radiation: Radiation Therapy
  Other Names: XRT
Drug: Temozolomide
  Other Names: temo; temodar
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
Studies which have separately studied bevacizumab for recurrent gliomas and bevacizumab for newly-diagnosed glioma have shown good results and the regimens have been well-tolerated by patients. This study seeks to investigate the use of bevacizumab with the standard therapy (radiation therapy and temozolomide) in newly diagnosed patients, followed by bevacizumab and temozolomide with the continuation of bevacizumab following progression. Two critical questions remain- the role of bevacizumab maintenance and bevacizumab at the time of progression in a patient previously treated with bevacizumab at the time of initial diagnosis.

DETAILED DESCRIPTION:
Given the possible synergism with irinotecan and bevacizumab for colorectal carcinomas, the combination has been studied in gliomas. In a study of 21 patients, the combination of irinotecan and bevacizumab produced a 43% response rate, with acceptable toxicity. The response rate is significantly higher than irinotecan alone and any other therapy for recurrent glioma. There were two serious adverse events, one intracranial hemorrhage and one bowel perforation. At the Duke Brain Tumor Center, the investigators have treated over 1000 glioblastoma patients with a bevacizumab-containing regimen, and there is marked clinical benefit and acceptable toxicity. Our initial study looking at the combination of bevacizumab and irinotecan for patients with recurrent glioblastoma published in 2007 found impressive response rates and survival and corroborated the earlier experience of Starks-Vance.

The investigators completed a study for newly diagnosed glioblastoma that utilized bevacizumab, radiation therapy and temozolomide followed by 6 months of bevacizumab, irinotecan and temozolomide. In addition, the group at University of California at Los Angeles published a study with bevacizumab, radiation therapy and temozolomide followed by 12 months of bevacizumab and temozolomide for newly diagnosed glioblastoma. These two phase II studies reported acceptable toxicity and a suggestion of improved survival compared to historical controls, and led to two large phase III randomized, placebo controlled studies of the addition of bevacizumab for newly diagnosed glioblastoma patients. The current proposal builds on the encouraging results of the addition of bevacizumab to the standard therapy for newly diagnosed glioblastoma patients. Two critical questions remain- the role of bevacizumab maintenance and bevacizumab at the time of progression in a patient previously treated with bevacizumab at the time of initial diagnosis. In addition, a retrospective analysis of data collected at our center from patients with recurrent disease suggests that continuation of bevacizumab at the time of progression may improve overall survival in comparison with cessation of bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed WHO Grade IV primary malignant glioma (glioblastoma or gliosarcoma);
* Patients ≥ 18 years of age;
* An interval of at least 2 weeks, but not ≥ 8 weeks between prior surgical procedure and initiation of treatment;
* Karnofsky Performance Status (KPS) ≥ 60%
* Laboratory Values:

  * Platelet Count ≥ 125,000 cells/µL
  * Absolute neutrophil count (ANC) ≥ 1,500 cells/µL
  * Adequate renal function indicated by all of the following:

    * Serum creatinine ≤ 1.25 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 ml/min
    * Urine dipstick for proteinuria < 2+ unless a 24-hour urine protein < 1 g of protein is demonstrated
  * internationalized normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤ 1.5 x upper limit of normal (ULN) within 7 days prior to first study treatment for patients not receiving anti-coagulation. The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least two weeks prior to the first study treatment.
* Patients will sign an Institutional Review Board-approved informed consent form.
* Female patients must not be pregnant or breast-feeding. Female patients of childbearing potential (defined as < 2 years after last menstruation or not surgically sterile) must use a highly effective contraceptive method (allowed methods of birth control, [i.e. with a failure rate of < 1% per year] are implants, injectables, combined oral contraceptives, intra-uterine device [Intrauterine Device (IUD); only hormonal], sexual abstinence or vasectomized partner) during the trial and for a period of > 6 months following the last administration of trial drug(s). Female patients with an intact uterus (unless amenorrhea for the last 24 months) must have a negative serum pregnancy test within 7 days prior to first study treatment.
* Fertile male patients must agree to use a highly effective contraceptive method (allowed methods of birth control [i.e. with a failure rate of < 1% per year] include a female partner using implants, injectables, combined oral contraceptives, Intrauterine Device (IUDs) [only hormonal], sexual abstinence or prior vasectomy) during the trial and for a period of > 6 months following the last administration of trial drugs.

Exclusion Criteria:

* Any prior treatment for any grade glioma, including, but not limited to gliadel wafers, immunotherapy (including vaccine therapy), radiation therapy or chemotherapy, irrespective of grade of the tumor (NOTE: 5-aminolevulinic acid (ALA)-mediated photodynamic therapy administered prior to surgery to aid in optimal surgical resection is not considered a chemotherapy agent.);
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids;
* Active infection requiring intravenous antibiotics;
* Prior or current treatment with bevacizumab or other anti-angiogenic treatment (i.e. anti-vascular endothelial growth factor (VEGF) or vascular endothelial growth factor receptor (VEGFR) therapies or tyrosine kinase inhibitors) for any condition;
* Treatment with any other investigational agent within 28 days or 2 investigational agent half-lives (whichever is longer) prior to first study treatment;
* Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin;
* Evidence of > Grade 1 central nervous system (CNS) hemorrhage on post-operative MRI scan, unless repeat MRI or CT performed prior to initiating bevacizumab shows stable grade 1 or resolving (< grade 1) CNS hemorrhage.

Bevacizumab-Specific Exclusion Criteria:

* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg) within 28 days of first study treatment;
* Prior history of hypertensive crisis, hypertensive encephalopathy, reverse posterior leukoencephalopathy syndrome (RPLS);
* Prior history of gastrointestinal perforation or abscess;
* Clinically significant (i.e. active) cardiovascular disease, for example cerebrovascular accidents ≤ 6 months prior to study enrollment, myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment;
* History or evidence upon physical/neurological examination of central nervous system disease (e.g. seizures) unrelated to cancer unless adequately controlled by medication or potentially interfering with protocol treatment;
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to start of study treatment. Any previous venous thromboembolism > NCI common toxicity criteria adverse event (CTCAE) Grade 3;
* History of pulmonary hemorrhage/hemoptysis ≥ grade 2 (defined as ≥ 2.5 mL bright red blood per episode) within 1 month of first study treatment;
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e. in the absence of therapeutic anticoagulation);
* Current or recent (within 10 days of study enrollment) use of aspirin (>325 mg/day), clopidogrel (>75 mg/day) or equivalent. Prophylactic use of anticoagulants is allowed;
* Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to first study treatment, or anticipation of need for major surgical procedure during the course of the study;
* Minor surgical procedure, e.g. stereotactic biopsy, within 7 days of first study treatment; placement of a vascular access device, within 2 days of first study treatment;
* History of intracranial abscess within 6 months prior to first study treatment;
* History of active gastrointestinal bleeding within 6 months prior to first study treatment;
* Serious, non-healing wound, active ulcer, or untreated bone fracture;
* Known hypersensitivity to any component of bevacizumab or any of the study drugs;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke Health
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

REFERENCES:
- See also: Preston Robert Tisch Brain Tumor Center at Duke — http://www.cancer.duke.edu/btc/
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/
- See also: Duke Cancer Center - Patient Care — http://www.dukehealth.org/cancer/locations/duke-cancer-center

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevaczimab, Radiation Therapy, Temozolomide: In Part A, newly-diagnosed patients with Grade 4 malignant gliomas will receive standard radiation therapy, daily Temodar 75mg/M for 6-8 weeks. Bevacizumab will be given concurrently with radiation therapy and Temodar, 10 mg/kg every two weeks.
  If they are stable at the end of Part A, they will continue to Part B. In Part B patients will receive up to 12 cycles of bevacizumab and Temodar. Bevacizumab will be given on Days 1 and 15 of a 28-day cycle. Temodar will be 200 mg/meter squared daily for 5 days (days 1-5) of each cycle.
  If they have not progressed, patients will start Part C. In Part C, patients will receive bevacizumab 10mg/kg approximately every 2 weeks or 15 mg/kg approximately every 3 weeks.
  If patients progress during Part B or C, they will start Part D. In Part D, patients will receive bevacizumab-based therapy containing bevacizumab in combination with a chemotherapy and/or biologic agent, as determined by the Duke treating physician.
  Radiation Therapy
  Temozolomide
  Bevacizumab
Period: Overall Study
Arm/Group | Bevaczimab, Radiation Therapy, Temozolomide
Started | 68
Entered Part A | 68
Entered Part B | 62
Entered Part C | 20
Entered Part D | 42
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevaczimab, Radiation Therapy, Temozolomide
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.43 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 64
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: To assess the effect on overall survival of continuing bevacizumab treatment after disease progression in patients treated with bevacizumab from the time of first diagnosis of grade IV malignant glioma.
Time Frame: 5 Years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevaczimab, Radiation Therapy, Temozolomide
Number analyzed (Participants) | 68
months | 17.8 [15.2 to 23.2]

2. Secondary Outcome: Toxicity: Percentage of Subjects With Unacceptable Toxicities
Description: The occurrence of ≥ grade 2 CNS (central nervous system) hemorrhage or grade 4 or 5 non-hematologic toxicity is defined as being unacceptable. "Unacceptable" toxicity rates of 5% or less are considered desirable, while rates of 20% or greater are considered as undesirable.
Time Frame: 5 Years
Measure: Number; unit: percentage of participants
Arm/Group | Bevaczimab, Radiation Therapy, Temozolomide
Number analyzed (Participants) | 68
percentage of participants | 11.8

3. Secondary Outcome: Progression-free Survival (PFS)
Description: To assess the effect on progression-free survival of continuing bevacizumab treatment after disease progression in patients treated with bevacizumab from the time of initiation of treatment to the first occurrence of progression, or death
Time Frame: 5 Years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevaczimab, Radiation Therapy, Temozolomide
Number analyzed (Participants) | 68
months | 9.9 [8.8 to 13.6]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Bevaczimab, Radiation Therapy, Temozolomide
All-Cause Mortality (participants affected / at risk) | 68/68
Serious Adverse Events (participants affected / at risk) | 41/68
Other Adverse Events (participants affected / at risk) | 68/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevaczimab, Radiation Therapy, Temozolomide (N=68)
Anemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Colonic perforation (Gastrointestinal disorders) | 1
Duodenal obstruction (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 8
Fatigue (General disorders) | 2
Fever (General disorders) | 5
Gait disturbance (General disorders) | 1
Localized edema (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Infections and infestations - Other, specify: R PERI-TONSILLAR ABSCESS; CPT-11 (Infections and infestations) | 1
Infections and infestations - Other, specify: ULCERATIVE VIRAL L TONSILLITIS (Infections and infestations) | 1
Infections and infestations - Other, specify: VIRAL SEPSIS SYNDROME (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Rash pustular (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 8
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Ataxia (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Intracranial hemorrhage (Nervous system disorders) | 1
Pyramidal tract syndrome (Nervous system disorders) | 6
Seizure (Nervous system disorders) | 15
Stroke (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 3
Proteinuria (Renal and urinary disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 7
Thromboembolic event (Vascular disorders) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevaczimab, Radiation Therapy, Temozolomide (N=68)
Anemia (Blood and lymphatic system disorders) | 45
Chest pain - cardiac (Cardiac disorders) | 1
Conduction disorder (Cardiac disorders) | 1
Mitral valve disease (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify: FULLNESS IN LEFT EAR-RADIATION (Ear and labyrinth disorders) | 1
Ear and labyrinth disorders - Other, specify: L EAR CLOGGED; XRT (Ear and labyrinth disorders) | 1
Ear and labyrinth disorders - Other, specify: WAX IMPACTION (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Endocrine disorders - Other, specify: HYPOTESTOSTERONEMIA (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 10
Cataract (Eye disorders) | 1
Dry eye (Eye disorders) | 2
Eye disorders - Other, specify: DIPLOPIA (Eye disorders) | 1
Eye disorders - Other, specify: EYE STRAIN (Eye disorders) | 1
Eye disorders - Other, specify: FLOATER VS. SMUDGE; XRT (Eye disorders) | 1
Eye disorders - Other, specify: HOMONYMOUS HEMIANOPSIA; RIGHT EYE (Eye disorders) | 1
Eye disorders - Other, specify: L EYE TWITCH FROM EYE STRAIN (Eye disorders) | 1
Eye disorders - Other, specify: L HOMONYMOUS HEMIANOPSIA (Eye disorders) | 2
Eye disorders - Other, specify: MOMENTARY LOSS OF VISION IN L EYE (Eye disorders) | 1
Eye disorders - Other, specify: OPTIC NERVE NEUROPATHY; AVASTIN (Eye disorders) | 1
Eye disorders - Other, specify: PERIPHERAL VISION LOSS (Eye disorders) | 1
Eye disorders - Other, specify: R VISUAL FIELD CUT (Eye disorders) | 1
Eye disorders - Other, specify: R VISUAL FIELD CUT, DISEASE PROGRESSION (Eye disorders) | 1
Eye disorders - Other, specify: RU QUADRANOPSIA (Eye disorders) | 2
Photophobia (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Anal hemorrhage (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 49
Dental caries (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 33
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 4
Fecal incontinence (Gastrointestinal disorders) | 7
Flatulence (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other, specify: ABSCESSED WISDOM TOOTH (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: CHIPPED TOOTH (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify: RECTAL BLEEDING; AVASTIN (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 2
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 5
Mucositis oral (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 42
Oral hemorrhage (Gastrointestinal disorders) | 3
Periodontal disease (Gastrointestinal disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 23
Chills (General disorders) | 1
Death NOS (General disorders) | 11
Edema limbs (General disorders) | 12
Fatigue (General disorders) | 63
Fever (General disorders) | 13
Flu like symptoms (General disorders) | 5
Gait disturbance (General disorders) | 4
Other, specify: DUE TO STEROIDS, INTERMITTENT DIAPHORESIS, LIGHTHEADEDNESS AND HYPERTENSION (General disorders) | 1
General disorders and administration site conditions - Other, specify: FEELS COLD (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Injection site reaction (General disorders) | 1
Irritability (General disorders) | 4
Localized edema (General disorders) | 1
Neck edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 10
Gallbladder obstruction (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 4
Bronchial infection (Infections and infestations) | 1
Infections and infestations - Other, specify: COLD SORES (Infections and infestations) | 1
Infections and infestations - Other, specify: GOUT (Infections and infestations) | 1
Infections and infestations - Other, specify: LYME'S DX (Infections and infestations) | 1
Infections and infestations - Other, specify: RLE CELLULITIS (Infections and infestations) | 1
Infections and infestations - Other, specify: SHINGLES (Infections and infestations) | 3
Infections and infestations - Other, specify: TRIGEMINAL HERPES ZOSTER (Infections and infestations) | 1
Infections and infestations - Other, specify: ULCERATIVE VIRAL L TONSILLITIS (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Lymph gland infection (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 11
Skin infection (Infections and infestations) | 4
Tooth infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 10
Vaginal infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 10
Fracture (Injury, poisoning and procedural complications) | 2
Injury, poisoning and procedural complications - Other, specify: ABDOMINAL BRUISING AT INJECTION (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify: BRUISING ON RIGHT THUMB (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify: HAND PUNCTURE (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 41
Alkaline phosphatase increased (Investigations) | 16
Aspartate aminotransferase increased (Investigations) | 37
Blood bilirubin increased (Investigations) | 18
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 18
Lymphocyte count decreased (Investigations) | 53
Neutrophil count decreased (Investigations) | 45
Platelet count decreased (Investigations) | 59
Weight gain (Investigations) | 2
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 51
Anorexia (Metabolism and nutrition disorders) | 18
Dehydration (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 60
Hyperkalemia (Metabolism and nutrition disorders) | 14
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 14
Hypoalbuminemia (Metabolism and nutrition disorders) | 29
Hypocalcemia (Metabolism and nutrition disorders) | 34
Hypoglycemia (Metabolism and nutrition disorders) | 22
Hypokalemia (Metabolism and nutrition disorders) | 31
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 37
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Metabolism and nutrition disorders - Other, specify: STEROID INDUCED DIABETES (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify: VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 30
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 5
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: ADHESIVE CAPSULITIS (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: BILATERAL LEG CRAMPING (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: CALF CRAMPS (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: HARD BONY SWELLING ON LEFT HEEL (Musculoskeletal and connective tissue disorders) | 1
Other, specify: INTERMITTENT PAIN IN R GROIN & CALF (Musculoskeletal and connective tissue disorders) | 1
Other, specify: L SHOULDER PARTIAL THICKNESS TEAR, BURSITIS (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: MUSCLE INJURY (Musculoskeletal and connective tissue disorders) | 1
Other, specify: PAIN FROM HISTORICAL SPORTS INJURIES IN EXTREMITIES (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: STEROID MYOPATHY (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Cognitive disturbance (Nervous system disorders) | 2
Concentration impairment (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 6
Dysarthria (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 19
Dysphasia (Nervous system disorders) | 17
Encephalopathy (Nervous system disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 4
Headache (Nervous system disorders) | 43
Hypersomnia (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 27
Nervous system disorders - Other, specify: ANOMIA (Nervous system disorders) | 1
Nervous system disorders - Other, specify: DYSMETRIA (Nervous system disorders) | 1
Nervous system disorders - Other, specify: GAIT UNSTEADINESS (Nervous system disorders) | 1
Nervous system disorders - Other, specify: PERIPHERAL NERVE COMPRESSION - R FOOT (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 14
Pyramidal tract syndrome (Nervous system disorders) | 17
Radiculitis (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 31
Sinus pain (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 7
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 6
Confusion (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 8
Hallucinations (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 11
Chronic kidney disease (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 5
Proteinuria (Renal and urinary disorders) | 46
Renal and urinary disorders - Other, specify: BLADDER PRESSURE (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify: BLADDER SPASMS (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 9
Urinary retention (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 2
Breast pain (Reproductive system and breast disorders) | 1
Dyspareunia (Reproductive system and breast disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: ABNORMAL PAP SMEAR (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: ATYPICAL DUCTAL HYPERPLASIA - LEFT BREAST (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 51
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 24
Dry skin (Skin and subcutaneous tissue disorders) | 13
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13
Skin and subcutaneous tissue disorders - Other, specify: BASAL CELL CARCINOMA REMOVAL (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: BILATERAL FOREARMS BRUISING, INTERMITTENT (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: BIOPSY OF SCAB IN SITU LEFT NOSE (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: CALLOUS PATCHES BILATERAL FEET (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: CALLUS-LIKE FORMATION ON FOOT SKIN GRAFTS (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: DELAYED WOUND HEALING; AVASTIN (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: ECZEMATOUS DERMATITIS L FOREARM (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: HIVES ON R FLANK - DUE TO STRESS (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: HIVES/RASH (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: HYPERPIGMENTED SKIN LESIONS; CARBOPLATIN (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: I&D OF MID-BACK BOIL (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: LACERATION REQUIRING SUTURES (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: LEFT LE SKIN LESION S/P PUNCH BIOPSY (Skin and subcutaneous tissue disorders) | 1
Other, specify: MILD ERYTHEMA AROUND THE RIGHT BACKSIDE WITH QUESTIONING RESOLVING IMPETIGO. (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: MULTIPLE ABRASIONS FROM FALL (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: NON-INFECTED INGROWN TOENAIL (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: PETECHIAE B/L THIGHS; AVASTIN (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: PIMPLE/BUG BITE (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: R AND L PLANTAR CALLUSES (Skin and subcutaneous tissue disorders) | 1
Other, specify: R HAND SMALL SKIN TEAR; SECONDARY TO LONG TERM STEROID USE (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: REDNESS FROM TICK BITE (Skin and subcutaneous tissue disorders) | 1
Other, specify: REDNESS/FLUSHING OF FACE; POSSIBLY DUE TO STEROIDS (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: SCALP FOLLICULITIS (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: SKIN TEAR/BRUISING LEFT ELBOW (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: SQUAMOUS CELL CARCINOMA ON NOSE (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Hematoma (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 39
Hypotension (Vascular disorders) | 3
Phlebitis (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 7
Vascular disorders - Other, specify: BILATERAL LE CLAUDICATION (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT01740258/Prot_SAP_000.pdf